CLINICAL TRIAL: NCT04562974
Title: Approche représentationnelle de l'Hippocampe Dans la Cognition : Étude en IRMf
Brief Title: Representational Approach to Hippocampal Functions : a fMRI Study
Acronym: SHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other); University Grenoble Alps (Other); Université Savoie Mont Blanc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A01592-37; 2020-A01592-37 (Other: ID RCB)
Record Dates: First submitted 2020-09-04; First posted 2020-09-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Memory, Episodic; Form Perception
Keywords: memory; neuropsychology; hippocampus; perception; neuroimaging
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group of 30 healthy subjects (Experimental): Perception and memory tasks inside a MRI-scanner for all participants
  Interventions: Device: MRI-scanner

INTERVENTIONS:
Device: MRI-scanner — Only one group of 30 participants is constituted. All participants will perform perception and memory tasks inside a MRI-scanner. Functional activity (BOLD signal) will be registered, as well as anatomical and behavioural data.

SUMMARY:
Although traditional neuropsychological models associate medial temporal lobe (MTL) regions to memory, and the hippocampus to episodic memory, there is growing evidence supporting an alternative view. The representational view of the MTL proposes that such regions depends on the representations processed rather than the cognitive processes. The aim of this project is to characterise the role played by MTL areas, and particularly the hippocampus, in mnemonic and non-mnemonic cognition. Hypotheses stemming from the representational view will thus be tested, using functional MRI among young healthy participants.

DETAILED DESCRIPTION:
Traditional neuropsychological models associate the medial temporal lobe (MTL) with episodic memory. Further, the hippocampus would be responsible for recollection, or the rich and contextualised retrieval of a memory; whereas the perirhinal cortex (PRC) would process familiarity, or the feeling that a stimulus has been encountered before, without remembering where or when it happened. However, there is growing evidence questioning this view, and supporting an alternative proposal. The representational view of the MTL proposes that such regions would not be organised according to cognitive processes, but rather according to the representations (or the mnemonic content, represented by a pattern of neuronal spikes. A 2018-fMRI study demonstrated that the engagement of the hippocampus in recollection depends on the presence of a spatial scene in the memory that is retrieved, and not on the reconstructive nature of the retrieval. However, this demonstration is incomplete, as the only process that was investigated is recollection. The current project aims to extend such results to memory processes such as familiarity, and even to non-mnemonic processes such as visual discrimination. A fMRI study will thus be conducted, where 30 healthy participants will first perform a visual-discrimination task on scenes and objects, before taking a recognition task, in which images will either be presented in full or in the form of circular cues only. Multivariate-Pattern Analyses (MVPA) will complete traditional fMRI analyses, in order to determine whether activity in the MTL can be categorised on the basis of representations through a machine-learning classifier.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to French Healthcare system
* No contraindication to MRI examination
* Age between 18 and 35 years-old
* Visual acuity permitting normal perception of stimuli or corrected sight

Exclusion Criteria:

* Existence of a pathology incompatible with the protocol : Heart, respiratory, haematological, caner, neurological disorder...
* Brain-modulating medical treatment
* Alcohol intake before examination
* Uncorrected visual disorder
* Cognitive deficit (criterion MMSE < 27)
* People protected by articles L1121-5 to L1121-8 of the CSP (pregnant women, under-18 subjects, people under judiciary or administrative surveillance)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Hippocampal activity during behavioural tasks in the MRI scanner | through study completion, an average of 1 year
  Activity will be recorded through the MRI whereas participants will perform the tasks. Outcome criteria consist in significant activity observed in participants hippocampus, depending on the experimental conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Moreaud, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

REFERENCES:
- [Result] Gardette J, Cousin E, Bourgin J, Torlay L, Pichat C, Moreaud O, Hot P. Hippocampal activity during memory and visual perception: The role of representational content. Cortex. 2022 Dec;157:14-29. doi: 10.1016/j.cortex.2022.09.004. Epub 2022 Sep 28. PMID 36272329